CLINICAL TRIAL: NCT05852262
Title: High-dose Cephalexin for Cellulitis (HI-DOCC)
Acronym: HI-DOCC
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Network of Canadian Emergency Researchers (NCER) (Unknown); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20230205-01T
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cellulitis
Keywords: Cellulitis; Cephalexin; Oral antibiotics; Treatment failure
MeSH Terms: conditions — Cellulitis | interventions — Cephalexin

STUDY DESIGN:
Intervention Model Description: The Investigators will conduct a parallel arm double-blind randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Eligible patients will be randomized (1:1) to high-dose versus standard-dose arms. The randomization sequence will be computer-generated by a statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose Cephalexin (Experimental): The intervention is high-dose cephalexin (1000mg PO QID) for seven days
  Interventions: Drug: Cephalexin
- Standard Dose Cephalexin (Active Comparator): The comparator is standard-dose cephalexin (500mg PO QID) plus oral placebo for seven days
  Interventions: Drug: Cephalexin

INTERVENTIONS:
Drug: Cephalexin — 1000 mg PO QID for 7 days
  Other Names: High-dose cephalexin
  Arms: High Dose Cephalexin
Drug: Cephalexin — 500 mg PO QID plus oral placebo for 7 days
  Other Names: Standard-dose cephalexin
  Arms: Standard Dose Cephalexin

SUMMARY:
Cellulitis is a common condition diagnosed and managed in the ED that carries significant burden on healthcare systems globally. Cellulitis is the 8th most common reason patients present to an ED in Canada. Among middle-aged patients (45-64 years) it is the 5th most common reason to visit an ED. This disease is responsible for significant healthcare system burden due to high hospitalization rates and subsequent costs. The Investigators conducted a health records review at two large urban EDs in Ottawa, and found that 29.6% of patients with cellulitis are admitted to hospital. In a separate study, The investigators found that the mean cost of care to hospitalize cellulitis patients for IV antibiotics was $10,145 CDN.

DETAILED DESCRIPTION:
Background Non-purulent cellulitis is a bacterial skin and soft tissue infection of the subcutaneous tissue. Group A streptococcus (Streptococcus pyogenes), beta-hemolytic streptococci and methicillin-susceptible Staphylococcus aureus are the most common bacteria causing non-purulent cellulitis. Patients typically present to the emergency department (ED) with pain, redness, swelling and induration (skin hardening due to inflammation) of the affected skin. A minority of patients may have fever or tachycardia. The diagnosis of cellulitis is clinical. Once the diagnosis is made, antibiotic treatment is initiated. The emergency physician must select the appropriate agent, oral versus intravenous (IV) route, dose, frequency and duration.

Rationale For ED adult patients with cellulitis, how does high-dose (1000 mg QID) cephalexin compare with standard-dose (500 mg QID) cephalexin with respect to antibiotic treatment failure, adverse events and health service utilization (i.e., need for IV antibiotics, unscheduled return ED visits and hospitalization)? Hypotheses (superiority): Treatment with high-dose cephalexin will lead to lower rates of oral antibiotic treatment failure than using standard-dose cephalexin.

Methods:

Study Design & Setting The investigators will conduct a multicentre, parallel-arm double-blind, individually randomized trial comparing high-dose (1000 mg) cephalexin to standard-dose (500 mg) cephalexin to treat ED adult patients with cellulitis. This is a superiority trial. The trial will be conducted at 8 Canadian EDs. A total sample size of 446 patients (223 per group) will be required.

Study Population Inclusion Criteria The Investigators will include adults (age ≥18 years) diagnosed with non-purulent cellulitis and determined by the treating emergency physician to be eligible for outpatient oral antibiotics.

Trial Intervention The study interventions are two accepted doses of oral cephalexin. The interventions will begin following randomization.

1. High-dose cephalexin. Patients randomized to this arm will receive a seven-day medication package of cephalexin 1000 mg (two 500 mg tablets per dose) to be taken four times daily. A duration of seven days was selected as this was the most common prescription duration in a survey of Canadian emergency physicians.32 The antibiotic pills will be provided in a dosette organized by dose and day.
2. Standard-dose cephalexin. Patients randomized to this arm will receive a seven-day medication package of cephalexin 500 mg (one 500 mg tablet and one placebo tablet per dose) to be taken four times daily.
3. Blinding. Both cephalexin and placebo will be encased in identical capsules, prepared and packaged independently by an external pharmacy. The patients, treating physician and research team (including outcome adjudicators) will be blinded.

Primary Outcome: Oral Antibiotic Treatment Failure The primary outcome is outpatient oral antibiotic treatment failure, defined as a change in antibiotic (change in class of oral antibiotic or step up to IV therapy) within 7 days due to worsening infection.

Secondary Outcomes

1. Clinical cure, defined as absence of treatment failure criteria, evaluated at day 8 and 30
2. Clinical response, defined as a reduction in lesion size ≥20% compared to baseline, evaluated at the day 3 and day 8 follow-up assessments
3. Unplanned visits to a healthcare provider (ED, family doctor) within 30 days
4. Unplanned hospitalization within 30 days.
5. Adverse events will be classified as serious or other and will be assessed at day 30 follow up. Serious adverse events will include anaphylaxis to study medication, development of Clostridium difficile colitis or unexpected deaths related to the infection or treatment. Other adverse events include nausea, vomiting, diarrhea, abdominal pain and rash.
6. Antibiotic intolerance, defined as change in treatment due to adverse events.
7. Antibiotic allergy, defined as change in treatment due to skin, respiratory, cardiovascular, or gastrointestinal symptoms requiring treatment with an antihistamine and/or epinephrine.
8. Medication adherence, with full adherence defined as patients who report taking all study medication over 7 days
9. Health-related quality of life measured using the EuroQoL-5D-5L36 instrument
10. Change in antibiotic treatment (oral or IV antibiotics) but does not meet worsening infection criteria (i.e., none of the following: new or persistent fever (temperature ≥38.0 °C), increasing area of erythema (in cm2) ≥20% from baseline, or increase in pain ≥2 points from baseline on the numeric rating scale), evaluated at 30 days.
11. Additional course of oral or IV antibiotics after 7 day course of oral cephalexin completed, evaluated at day 30.
12. Recurrence of infection at day 30, defined as initially having met clinical cure criteria at day 3 or 8, but then developed a subsequent recurrent cellulitis within 30 days.

IMPORTANCE Cellulitis is a common cause of ED visits, and many patients are hospitalized. Current evidence is lacking regarding the optimal management of cellulitis. If high-dose cephalexin is found to be superior to standard-dose cephalexin, this will change practice, with the potential to reduce unnecessary IV antibiotic use, hospitalization, and costs. The results will help inform future skin and soft tissue infection treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

Adults (age ≥18 years) diagnosed with non-purulent cellulitis and determined by the treating emergency physician to be eligible for outpatient oral antibiotics.

Exclusion Criteria:

1. Age <18 years;
2. Patient already taking oral antibiotics;
3. Treating physician decides IV antibiotics are required;
4. Abscess requiring an incision and drainage procedure;
5. Known prior skin or soft tissue infection secondary to methicillin-resistant Staphylococcus aureus (MRSA);
6. Cellulitis secondary to a human or animal bite wound;
7. Penetrating wound or water exposure resulting in cellulitis;
8. Surgical site infection;
9. Patient found at a follow up visit to have an alternative, non-infectious etiology (e.g., deep vein thrombosis);
10. bilateral symptoms (e.g., both legs involved);
11. Malignancy and currently being treated with chemotherapy;
12. Solid organ or bone marrow transplant recipient;
13. Renal impairment with an estimated glomerular filtration rate <30 mL/min documented on the health record at any time within the past three months;
14. Allergy to cephalosporins or history of anaphylaxis to penicillin;
15. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Oral Antibiotic Treatment Failure | 7 days
  defined as a change in antibiotic (change in class of oral antibiotic or step up to IV therapy) within 7 days due to worsening infection. Any of the following meet criteria for worsening infection (at day 3 or 8 follow-up): (1) New fever (temperature ≥38.0C) or persistent fever at follow-up; (2) Increasing area of erythema (in cm2) ≥20% from baseline; or (3) Increasing pain ≥2 points from baseline (using the numeric rating scale).

SECONDARY OUTCOMES:
Number of Participants with clinical cure | evaluated at day 8 and day 30
  defined as absence of pain, erythema, and fever
Number of Participants with clinical response | evaluated at days 3 and 8
  defined as a reduction in lesion size ≥20% compared to baseline
Number of Participants with unplanned visits to a healthcare provider for cellulitis | 30 days
Number of Participants with unplanned hospitalization for cellulitis | 30 days
Number of Participants with adverse events | 30 days
  classified as serious or other and will be assessed at day 30 follow up. Serious adverse events will include anaphylaxis to study medication, development of Clostridium difficile colitis or unexpected deaths related to the infection or treatment. Other adverse events include nausea, vomiting, diarrhea, abdominal pain and rash.
Number of Participants with antibiotic intolerance | 7 days
  defined as change in treatment due to adverse events
Number of Participants with antibiotic allergy | 7 days
  defined as change in treatment due to skin, respiratory, cardiovascular, or gastrointestinal symptoms requiring treatment with an antihistamine and/or epinephrine.
Number of Participants with medication adherence | 7 days
  with full adherence defined as patients who report taking all study medication over 7 days
Number of Participants with health-related quality of life | 30 days
  Measured using EuroQol-5D-5L instrument at index visit and all follow-ups (days 3,8 and 30)
Change in antibiotic but not meeting worsening infection | Evaluated at 30 days
  Number of patients that had a change in antibiotic treatment (oral or IV antibiotics) but did not meet worsening infection criteria (i.e., none of the following: new or persistent fever (temperature ≥38.0 °C), increasing area of erythema (in cm2) ≥20% from baseline, or increase in pain ≥2 points from baseline on the numeric rating scale)
Additional antibiotics | Evaluated at 30 days
  Number of patients that received an additional course of oral or IV antibiotics after 7 day course of oral cephalexin completed
Recurrence | Evaluated at 30 days
  Number of patients that had a recurrence of infection at day 30, defined as initially having met clinical cure criteria at day 3 or 8, but then developed a subsequent recurrent cellulitis

CONTACTS AND LOCATIONS:
Overall Officials: Krishan Yadav, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (10):
- Canada (10):
  - South Health Campus, Calgary, Alberta
  - Queen Elisabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Thunder Bay Health Sciences Centre, Thunder Bay, Ontario
  - Sinai Health System, Toronto, Ontario
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Enfant-Jésus Hospital, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No